CLINICAL TRIAL: NCT04419129
Title: Department of Orthopedics, Faculty of Medicine, Thammasat University
Brief Title: Comparison of Functional Recovery Between Mobile Bearing Unicompartmental Knee Arthroplasty and Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Boonchana Pongcharoen, Associate Professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ThmmasatU
Record Dates: First submitted 2017-05-28; First posted 2020-06-05 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Patient Reported Outcome Measure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile bearing unicompartmental knee arthroplasty (Active Comparator): 50 mobile bearing UKA
  Interventions: Device: Oxford UKA
- posterior stabilized fixed bearing total knee arthroplasty (Active Comparator): 50 posterior stabilized fixed bearing cemented total knee arthroplasty
  Interventions: Device: Vanguard TKA

INTERVENTIONS:
Device: Oxford UKA — knee arthroplasty
  Arms: Mobile bearing unicompartmental knee arthroplasty
Device: Vanguard TKA — knee arthroplasty
  Arms: posterior stabilized fixed bearing total knee arthroplasty

SUMMARY:
The total knee replacement (TKA) has shown excellent survival. However, some patients were up to 20%, they still had pain and make them dissatisfy after operation. The medial unicompartmental knee arthroplasty (UKA) also has shown excellent survivorship. The patient who underwent UKA fell like normal knee because restoring natural kinematic and biomechanic compare to TKA. However, The previous studies did not include the same characteristic of patient in their studies. Therefor, UKA should be better than TKA. This study will compare TKA to mobile bearing medial UKA or Oxford medial UKA. The mobile bearing UKA is different to fixed bearing UKA. The mobile bearing UKA will be back knee alignment to pre-disease stage, restore knee stability and restore natural knee kinematic and biomechanic. Therefore, patients who underwent mobile bearing UKA will feel like normal knee and restore function to near or nearly normal. The measurement of clinical outcome after knee arthroplasty is questionable. The self-report questionnaire was used in the past. However, this score can not estimate the true function of patients. The patient have shown high score, but they still had pain and did not show satisfy after operation.The performance-based test such as 2-minute walk test (2MWT), 6-minute walk test (6MWT) and Timed get-up-and-go test (TUG) should show the exactly clinical outcome of patient following knee arthroplasty compare to self-report questionnaire. Today, no randomized controlled trial study to compare performance-based test between TKA and mobile bearing UKA. Therefor, this study will compare 2MWT and TUG between TKA and mobile bearing UKA in medial OA knee.

DETAILED DESCRIPTION:
The inclusion criteria were patients with medial of the knee with an Alhback score of 2, 3 or 4, those who were older than 40 years of age, those with a range of motion (ROM) > 90°, those with a varus deformity < 25°, and those with a flexion contracture < 20°. They were randomized into 2 groups using computer program. Group I was 50 UKAs and group II was 50 TKAs. All patients in group I received medial mobile-bearing UKA (Oxford® UKA; Zimmer Biomet, Inc, Warsaw, IN, USA) and group II received posterior stabilized fixed bearing total knee arthroplasty (Vanguard®; Zimmer Biomet, Inc, Warsaw, IN, USA). The exclusion criteria were patients with a diagnosis of spontaneous osteonecrosis of the knee (SPONK), intraoperative anterior cruciate ligament (ACL) insufficiency or completely rupture of ACL, inflammatory joint disease, gout, posttraumatic arthritis, or primary patellofemoral arthritis.The recorded baseline patient characteristics included age and sex and the knee side, Knee Society Score (KSS), Oxford Knee Score (OKS), Knee Injury and Osteoarthritis Outcome Score (KOOS),(2MWT), (6MWT), (TUG), body mass index (BMI), degree of varus deformity, degree of flexion contracture, genu recurvatum, and ROM. Patients were followed at 6 weeks, 3 months, 6 months, and 1 year and then annually thereafter. At each follow-up, the following data were recorded: Joint Forgotten Score (JFS), KSS, OKS, Knee Injury and Osteoarthritis Outcome Score (KOOS), Kujala score, (2MWT), (TUG), ROM and knee alignment. In addition, the following knee X-rays were performed: anteroposterior (AP) and lateral standing, skyline and long-leg views; from these, the tibiofemoral angles were measured. Complications such as infection, component loosening, fractures, and bearing dislocations were also recorded. We determined differences in the KSS, OKS, KOOS, JFS, Kujala score,(2MWT), (TUG),ROM, tibiofemoral angle, flexion contractures, and genu recurvatum using Student's t tests. All analyses were two sided, and a p value of ≤ 0.05 denoted statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* anteromedial OA knee

Exclusion Criteria:

* varus deformity > 15 degrees
* ROM < 90 degrees
* fixed varus deformity
* post-traumatic arthritis
* inflammatory arthritis
* anterior cruciate ligament insufficiency

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
2 minutes walk test (2MWT) | 2 years
  measurement of endurance that assesses walking distance over 2 minutes
time up and go test (TUG) | 2 years
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.

SECONDARY OUTCOMES:
Knee Society Score | 2 years
  The standard clinical evaluation system for reporting results for patients undergoing unicompartmental knee arthroplasty
Oxford knee score | 2 years
  The standard clinical evaluation system for reporting results for patients undergoing unicompartmental knee arthroplasty
Forgotten Joint Score | 2 years
  The standard clinical evaluation system for reporting results for patients undergoing unicompartmental knee arthroplasty
Kujala score | 2 years
  The standard clinical evaluation system for reporting results for patients undergoing unicompartmental knee arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Boonchana Pongcharoen, MD, Study Director — faculty of medicine, Thammasat university
Locations (1):
- Boonchana Pongcharoen, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pongcharoen B, Liengwattanakol P, Boontanapibul K. Comparison of Functional Recovery Between Unicompartmental and Total Knee Arthroplasty: A Randomized Controlled Trial. J Bone Joint Surg Am. 2023 Feb 1;105(3):191-201. doi: 10.2106/JBJS.21.00950. Epub 2022 Dec 21. PMID 36542689